CLINICAL TRIAL: NCT04918745
Title: VertiGO! - Get up and GO! With the Vestibular Implant
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: University Hospital, Geneva (Other); MED-EL Elektromedizinische Geräte GesmbH (Industry); Health Holland (Other); Heinsius-Houbolt Fund (Unknown); Radboud University Medical Center (Other); Stichting de Weijerhorst (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: NL73492.068.20; METC20-087 (Other: METC azM/UM)
Record Dates: First submitted 2021-04-28; First posted 2021-06-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Bilateral Vestibular Loss
Keywords: Vestibular Implant; Cochlear vestibular implant; Bilateral vestibulopathy; Bilateral vestibular hypofunction; Bilateral vestibular loss; Cochlear implant
MeSH Terms: conditions — Bilateral Vestibulopathy

STUDY DESIGN:
Intervention Model Description: Controlled clinical trial with a randomized single-blind 3-treatment 3-period crossover design during the in-hospital part
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- ABC (Other): In-hospital part
  A = Baseline stimulation, no modulation
  B = Baseline stimulation, modulation stimulation
  C = Reduced baseline stimulation, modulation stimulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)
- ACB (Other): In-hospital part
  A = Baseline stimulation, no modulation
  C = Reduced baseline stimulation, modulation stimulation
  B = Baseline stimulation, modulation stimulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)
- BAC (Other): In-hospital part
  B = Baseline stimulation, modulation stimulation
  A = Baseline stimulation, no modulation
  C = Reduced baseline stimulation, modulation stimulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)
- BCA (Other): In-hospital part
  B = Baseline stimulation, modulation stimulation
  C = Reduced baseline stimulation, modulation stimulation
  A = Baseline stimulation, no modulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)
- CAB (Other): In-hospital part
  C = Reduced baseline stimulation, modulation stimulation
  A = Baseline stimulation, no modulation
  B = Baseline stimulation, modulation stimulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)
- CBA (Other): In-hospital part
  C = Reduced baseline stimulation, modulation stimulation
  B = Baseline stimulation, modulation stimulation
  A = Baseline stimulation, no modulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)
- 1122 (Other): Home-use part, preference phase
  1. - individualized vestibular stimulation
  2. - control vestibular stimulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)
- 1212 (Other): Home-use part, preference phase
  1. - individualized vestibular stimulation
  2. - control vestibular stimulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)
- 1221 (Other): Home-use part, preference phase
  1. - individualized vestibular stimulation
  2. - control vestibular stimulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)
- 2211 (Other): Home-use part, preference phase
  1. - individualized vestibular stimulation
  2. - control vestibular stimulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)
- 2121 (Other): Home-use part, preference phase
  1. - individualized vestibular stimulation
  2. - control vestibular stimulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)
- 2112 (Other): Home-use part, preference phase
  1. - individualized vestibular stimulation
  2. - control vestibular stimulation
  Interventions: Device: Cochlear Vestibular Implant (CVI)

INTERVENTIONS:
Device: Cochlear Vestibular Implant (CVI) — The Cochlear Vestibular Implant (CVI) is a modified cochlear implant (CI) which also incorporates a vestibular component (VI) in order to restore both hearing and vestibular function.
  During the in-hospital part, three vestibular stimulation algorithms will be compared in a randomized order (3 treatments x 3 periods, = 6 arms). These stimulation algorithms are:
  * A - Baseline stimulation, no modulation stimulation
  * B - Baseline stimulation, modulated stimulation
  * C - Reduced baseline stimulation, modulated stimulation
  During the home-use part, a preference phase will be included to assess the effects of a "control". Participants will receive two research processors, each with a different vestibular stimulation mode. These modes will be randomized over a 4-week period, each appearing twice (2 treatments appearing twice each x 4 weeks = 6 arms). These stimulation modes are:
  * 1 - individualized vestibular stimulation
  * 2 - control vestibular stimulation

SUMMARY:
In the VertiGO! trial 13 participants with bilateral vestibulopathy (BV) and severe sensory neural hearing loss in the ear to be implanted will receive a combined cochlear (CI) and vestibular implant (VI), capable of stimulating both the cochlear and vestibular nerves (CVI). The participants will firstly make use of this combined stimulation during 3 weeks of prolonged use under direct supervision in a hospital environment. Following this, participants will make use of combined stimulation in a real-life environment (e.g., outside of the hospital setting) for 15 months under indirect supervision. This trial will serve as a proof-of-concept for restoring vestibular function in patients with BV, an as-of-yet untreatable disorder causing severe impairment and discomfort. The aims of this trial are to investigate efficacy and safety of prolonged vestibular stimulation, to identify the influence of different stimulation algorithms, to assess the feasibility of the combined VI/CI device, to develop a VI rehabilitation program and to further build on the fundamental knowledge of vestibular organ stimulation while also taking into account the patient perspective.

DETAILED DESCRIPTION:
The vestibular sensory organ is essential for balance and image stabilization. Patients with severe function loss of both vestibular organs present themselves with serious day-to-day disabilities such as strong balance disturbances, higher risk of falling, visual symptoms (oscillopsia) and a loss of autonomy. Up until now no effective treatment is available for these patients to restore vestibular function. In the past years experimental electric stimulation of the vestibular nerve in humans by means of a VI has shown to be able to partly restore balance and gaze functionality in test situations.

To evaluate combined prolonged stimulation of both the vestibular organ and the cochlea, participants will be implanted with a CVI. This modified CI also consists of 3 vestibular electrodes, each placed in individual electrode leads for insertion into the three semicircular canals. Therefore the CVI is capable of stimulating both the cochlear and vestibular nerves. Hearing rehabilitation with the CI part of the device will follow the standard clinical protocol, with the participant using a standard CI processor. Functionality of prolonged combined vestibular and cochlear stimulation will first be assessed using a research processor during 3 weeks (3x4 days, +- 8 hours a day) of prolonged stimulation under direct supervision in the safety of a hospital environment. This is considered the in-hospital part. Following this, a modified research processor will be used during 15 months (13 visits, half and full day) of prolonged stimulation in real-life situations under indirect supervision. This is considered the home-use part of the trial.

During the in-hospital part, each identical period of 4 days a different stimulation algorithm will be used for vestibular stimulation, with the order being randomized and single-blinded. The stimulation algorithms which will be used are (1) baseline stimulation without motion modulation, (2) baseline stimulation with motion modulation, and (3) reduced baseline stimulation with motion modulation.

During the home-use part, the efficacy and safety of prolonged VI stimulation will be evaluated in a home environment using pre-post intervention evaluation. During this part, the stimulation status will alternate between VI-ON and VI-OFF, depending on the phase. The stimulation algorithm will be optimized per patients to best evaluate VI efficacy (optimization phase). Furthermore, safety and efficacy will be further elucidated by maintaining consistent prolonged VI stimulation (persistency phase), using a consistent algorithm with minimal adjustments. Following this, a resting period of at least four weeks (washout phase) will commence, where no VI stimulation will be used. This will allow for comparison between vestibular stimulation (VI-ON) versus without stimulation (VI-OFF), which aligns with the primary comparison used during the in-hospital period. In addition, this phase aims to minimize carry-over effect, ensure adequate resolution of aftereffects and evaluation of changes to quality of life. Finally, evaluation of single blinded preference between stimulation statuses will be assessed (preference phase). Patients will have the option to continue using vestibular stimulation after the preference phase for as long as the trial continues (resume phase).

Alongside the periods of prolonged stimulation, the participant will make yearly visits to our clinic up to 5 years after implantation for evaluation of long-term response to acute vestibular stimulation and general CI performance.

ELIGIBILITY:
Inclusion criteria:

1. Chronic vestibular syndrome being presented by disabling symptoms of postural imbalance and/or impaired image stabilization (e.g. oscillopsia)
2. Reduced or absent bilateral VOR function based on at least one of the tests below meeting criteria A, with the other tests meeting criteria B:

   Criteria A: Caloric response: Each side ≤6°/sec, vHIT gain: Bilateral horizontal SCC ≤ 0.6 AND Bilateral vertical SCC <0.7, Rotatory chair gain: ≤ 0.1 (0.1 Hz)

   Criteria B: Caloric response: Each side <10°/sec, vHIT gain: 2 Bilateral SCC <0.7, Rotatory chair gain: ≤ 0.2 (0.1 Hz)
3. Onset of bilateral vestibular loss after the age of 2
4. Vestibular dysfunction from a peripheral origin or idiopathic BV
5. Patent vestibular end-organ (judged by CT)
6. Vestibular function and symptoms have not recovered beyond inclusion criteria within 6 months from onset of symptoms including a 3 month rehabilitation program off vestibular suppressant medications
7. Meeting CI-candidacy in ear to implant with CVI
8. Agreed to receive a MED-EL CVI implant with MED-EL sound processor
9. Capacitated adults ≥ 18 years
10. Proficient speaker of the Dutch language
11. No contra-indications for CVI surgery
12. Active participation in the trial related procedures such as regular testing, the VI fitting period, the baseline testing day and three weeks of intensive VI rehabilitation and testing in the study center (MUMC+) including an exercise regimen
13. Agreed not to swim or to use or operate vehicles, heavy machinery, powered tools or other devices that could pose a threat to the participant, to others, or to property throughout the period of VI activation and until at least 1 day after VI deactivation

Remark: Patients who qualify to receive a regular CI as part of standard clinical care will have a preferential position to be included in the trial.

Exclusion Criteria:

1. Signs of central vestibular/cochlear dysfunction or structural vestibular/cochlear nerve pathology (judged by physical examination / MRI)
2. Clear signs of structural nerve pathology or indications of improperly functioning vestibular/cochlear nerves
3. Requirement for electric-acoustic activation of the CI part (e.g. "hybrid" processor) prior to completion of the prolonged VI stimulation period
4. Having received a cochlear implant earlier on the side to implant (e.g. explantation/reimplantation)
5. Having received a cochlear implant from another brand than MED-EL in the other ear (bilateral implantation with different brands is not supported)
6. Unwillingness to stop the use of antihistamines which might suppress VOR responses (e.g. cinnarizine) in the period of 1 month before until after each measurement point.
7. Pre-lingual onset of bilateral profound deafness (< 4 years of age)
8. Active participation in another prospective clinical trial
9. Pregnancy or having plans to become pregnant at the time of imaging or during the VI trial
10. Orthopedic, ocular, neurologic or other non-vestibular pathologic conditions of sufficient severity to confound vestibular function tests used in the study
11. Current psychological or psychiatric disorders that could significantly interfere with the use or evaluation of VI stimulation
12. Physical or non-physical contraindications for MRI or CT imaging prior to surgery
13. Making chronic use of psychiatric medication which suppresses VOR responses (e.g. SSRI's, benzodiazepines)
14. Significant dental problems which prohibit the stable use of a 'bite bar' (used as calibration reference for the gyroscope functionality of the CVI)
15. Any medical condition, judged by the research team, that is likely to interfere with a study candidate's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of vestibular stimulation via the CVI | Through full trial period, up to 5 years postoperatively
  Amount of (S)AE's after implantation to determine safety of the device
The feasibility of vestibular stimulation improving Dynamic Visual Acuity during walking | Through all stimulation periods, within 5 years after implantation
  Quantifying vestibulo-ocular reflex restoration on a functional level by evaluating the capacity of vestibular stimulation (via the CVI) to improve dynamic visual acuity while walking. Adaptation to vestibular stimulation will be evaluated through the in-hospital and home-use parts.
The feasibility of vestibular stimulation improving Dynamic Visual Acuity during passive head movements | Through each 4-day VI stimulation period, within 2 years after implantation
  Quantifying vestibulo-ocular reflex restoration on a functional level by evaluating the capacity of vestibular stimulation (via the CVI) to improve dynamic visual acuity during fast passive head movements measured with the functional Head Impulse Test. Adaptation to stimulation will be evaluated through each 4-day stimulation period with each stimulation algorithm being evaluated separately.
The feasibility of vestibular stimulation restoring the high-frequency vestibulo-ocular reflex | Through each 4-day VI stimulation period, within 2 years after implantation
  Evaluating the capacity of vestibular stimulation (via the CVI) to increase vestibulo-ocular reflex gain during fast passive head movements in the LHRH, RALP and LARP planes measured with the video Head Impulse Test. Adaptation to stimulation will be evaluated through each 4-day stimulation period with each stimulation algorithm being evaluated separately.
The feasibility of vestibular stimulation restoring the low-frequency vestibulo-ocular reflex | Through each 4-day VI stimulation period, within 2 years after implantation
  Evaluating the capacity of vestibular stimulation (via the CVI) to increase vestibulo-ocular reflex gain during slow, passive, full body rotations measured with the Torsion Swing test. Adaptation to stimulation will be evaluated through each 4-day stimulation period with each stimulation algorithm being evaluated separately.
The feasibility of vestibular stimulation improving the self-movement perception in dark | Through each 4-day VI stimulation period, within 2 years after implantation
  Evaluating whether vestibular stimulation (via the CVI) can improve self-motion perception measured by controlled motion stimuli delivered by a moving platform. Adaptation to stimulation will be evaluated through each 4-day stimulation period with each stimulation algorithm being evaluated separately.
The feasibility of vestibular stimulation improving gait stability and balance based on motion capture data on a treadmill | Through each 4-day VI stimulation period, within 2 years after implantation
  Evaluating the influence of vestibular stimulation (via the CVI) on walking patterns and stability based on motion capture data. Adaptation to stimulation will be evaluated through each 4-day stimulation period with each stimulation algorithm being evaluated separately.
The feasibility of vestibular stimulation improving gait stability and balance based on motion capture data overground | Through each home-use phase, within 5 years after implantation
  Evaluating the influence of vestibular stimulation (via the CVI) on walking patterns and stability based on motion capture data. Adaptation to vestibular stimulation will be evaluated through each phase during the home-use part of the trial.
The feasibility of vestibular stimulation improving balance based on clinical evaluation | Through each 4-day VI stimulation period, within 2 years after implantation
  Clinical evaluation of the influence of vestibular stimulation (via the CVI) on balance measured with the MiniBESTest. Adaptation to stimulation will be evaluated through each 4-day stimulation period with each stimulation algorithm being evaluated separately.
Speech perception with CVI in quiet without simultaneous vestibular stimulation | Through the full trial period, until 5 years after implantation
  Evaluating hearing performance with the CVI based on speech perception in quiet measured with an aided consonant-nucleus-consonant word test, without simultaneous vestibular stimulation
Interaction between vestibular and cochlear stimulation on speech perception in quiet | Through each 4-day VI stimulation period, within 2 years after implantation
  Evaluating hearing performance with the CVI based on speech perception in quiet while simultaneously providing vestibular stimulation, measured with an aided consonant-nucleus-consonant word test. The influence of each vestibular stimulation algorithm will be evaluated separately.
Speech perception with CVI in noise without simultaneous vestibular stimulation | Through the full trial period, until 5 years after implantation
  Evaluating hearing performance with the CVI based on speech perception in noise measured with a sentence speech In noise test, without simultaneous vestibular stimulation
Change in otolith function due to CVI implantation | preoperatively and 1 month postoperatively
  Evaluating the influence of CVI implantation on otolith function based on cVEMP and oVEMP responses post-operatively, comparing with the pre-operative situation.
Vestibular and cochlear electrode location | Through the full trial period, until 5 years after implantation
  Evaluating the location and potential migration of the vestibular and cochlear electrodes of the CVI with cone-beam CT scans- of the mastoid.

SECONDARY OUTCOMES:
Characterization of study population on perceived dizziness | Measured pre-operatively and directly before the start of the VI stimulation period
  Characterizing the study population based on their perceived dizziness and the related handicap measured with the Dizziness Handicap Inventory.
Characterization of study population on perceived risk of falling | Measured pre-operatively and directly before the start of the VI stimulation period
  Characterizing the study population based on their perceived risk of falling measured with the Falls Efficacy Scale-International
Characterization of study population on perceived severity of oscillopsia | Measured pre-operatively and directly before the start of the VI stimulation period
  Characterizing the study population based on their perceived severity of oscillopsia measured with the Oscillopsia Severity Questionnaire
Subjective hearing performance of the CVI | Yearly evaluation through the full trial period, until 5 years after implantation
  Evaluating the subjective hearing performance of the CVI measured with the Speech and Spatial Qualities of hearing scale-12
Effect of CVI implantation on tinnitus burden | Pre-operatively and 1 month postoperatively
  Evaluating the influence of CVI implantation on the subjective severity and burden of tinnitus measured with the Tinnitus Questionnaire
Characterization of study population on perceived health-related quality of life | Measured pre-operatively and directly before the start of the VI stimulation period
  Characterizing the study population based on their perceived health-related quality of life measured with the Health Utility Index - 3
Evaluating the influence of receiving and using a CVI on quality of life | Through the full trial period, until 5 years after implantation
  Evaluating the influence of the different stages of receiving and using a CVI on quality of life measured with the EuroQOL 5 Dimensional questionnaire. Aimed at separating CI-only use and full CVI use throughout the trial to get an accurate assessment of the influence vestibulo-cochlear electrical stimulation (via the CVI) can have on quality of life
Evaluating the influence of receiving and using a CVI on capabilities in life | Through the full trial period, until 5 years after implantation
  Evaluating the influence of the different stages of receiving and using a CVI on capabilities in life measured with the ICEPOP Capability measure for adults. Aimed at separating CI-only use and full CVI use throughout the trial to get an accurate assessment of the influence vestibulo-cochlear electrical stimulation (via the CVI) can have on quality of life.
Evaluating the influence of receiving and using a CVI on anxiety and depression | Through the full trial period, until 5 years after implantation
  Evaluating the influence of the different stages of receiving and using a CVI on anxiety and depression measured with the Hospital Anxiety and Depression Scale. Aimed at separating CI-only use and full CVI use throughout the trial to get an accurate assessment of the influence vestibulo-cochlear electrical stimulation (via the CVI) can have on these aspects.
Evaluating the daily experience with vestibular stimulation | Through each 4-day VI stimulation period, within 2 years after implantation
  A self-developed visual-analog scale-based list of questions for evaluating the participant's experience with the CVI on a daily basis during the prolonged stimulation period.
Characterizing the participant's experience with vestibular stimulation | Through each 4-day VI stimulation period, within 2 years after implantation
  Semi-standardized interviews for in-depth qualitative analysis of the participant's experience with receiving vestibular stimulation (via the CVI)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond van de Berg, MD, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized data will be shared via scientific publications in open source, peer-reviewed journals. Pseudonymized data will also be available upon request (see below).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 6 months after completion of the prolonged stimulation period
Access Criteria: A data agreement including research proposal needs to be signed prior to data sharing.

REFERENCES:
- [Background] Wall C 3rd, Kos MI, Guyot JP. Eye movements in response to electric stimulation of the human posterior ampullary nerve. Ann Otol Rhinol Laryngol. 2007 May;116(5):369-74. doi: 10.1177/000348940711600509. PMID 17561766
- [Background] van de Berg R, Guinand N, Stokroos RJ, Guyot JP, Kingma H. The vestibular implant: quo vadis? Front Neurol. 2011 Aug 11;2:47. doi: 10.3389/fneur.2011.00047. eCollection 2011. PMID 21991260
- [Background] Guyot JP, Sigrist A, Pelizzone M, Kos MI. Adaptation to steady-state electrical stimulation of the vestibular system in humans. Ann Otol Rhinol Laryngol. 2011 Mar;120(3):143-9. doi: 10.1177/000348941112000301. PMID 21510138
- [Background] van de Berg R, Guinand N, Guyot JP, Kingma H, Stokroos RJ. The modified ampullar approach for vestibular implant surgery: feasibility and its first application in a human with a long-term vestibular loss. Front Neurol. 2012 Feb 20;3:18. doi: 10.3389/fneur.2012.00018. eCollection 2012. PMID 22363317
- [Background] Perez Fornos A, Guinand N, van de Berg R, Stokroos R, Micera S, Kingma H, Pelizzone M, Guyot JP. Artificial balance: restoration of the vestibulo-ocular reflex in humans with a prototype vestibular neuroprosthesis. Front Neurol. 2014 Apr 29;5:66. doi: 10.3389/fneur.2014.00066. eCollection 2014. PMID 24808890
- [Background] Nguyen TA, Ranieri M, DiGiovanna J, Peter O, Genovese V, Perez Fornos A, Micera S. A real-time research platform to study vestibular implants with gyroscopic inputs in vestibular deficient subjects. IEEE Trans Biomed Circuits Syst. 2014 Aug;8(4):474-84. doi: 10.1109/TBCAS.2013.2290089. PMID 25073124
- [Background] Pelizzone M, Fornos AP, Guinand N, van de Berg R, Kos I, Stokroos R, Kingma H, Guyot JP. First functional rehabilitation via vestibular implants. Cochlear Implants Int. 2014 May;15 Suppl 1:S62-4. doi: 10.1179/1467010014Z.000000000165. No abstract available. PMID 24869447
- [Background] van de Berg R, van Tilburg M, Kingma H. Bilateral Vestibular Hypofunction: Challenges in Establishing the Diagnosis in Adults. ORL J Otorhinolaryngol Relat Spec. 2015;77(4):197-218. doi: 10.1159/000433549. Epub 2015 Sep 15. PMID 26366566
- [Background] van de Berg R, Guinand N, Nguyen TA, Ranieri M, Cavuscens S, Guyot JP, Stokroos R, Kingma H, Perez-Fornos A. The vestibular implant: frequency-dependency of the electrically evoked vestibulo-ocular reflex in humans. Front Syst Neurosci. 2015 Jan 20;8:255. doi: 10.3389/fnsys.2014.00255. eCollection 2014. PMID 25653601
- [Background] Guinand N, van de Berg R, Cavuscens S, Stokroos RJ, Ranieri M, Pelizzone M, Kingma H, Guyot JP, Perez-Fornos A. Vestibular Implants: 8 Years of Experience with Electrical Stimulation of the Vestibular Nerve in 11 Patients with Bilateral Vestibular Loss. ORL J Otorhinolaryngol Relat Spec. 2015;77(4):227-240. doi: 10.1159/000433554. Epub 2015 Sep 15. PMID 26367113
- [Background] Guinand N, van de Berg R, Ranieri M, Cavuscens S, DiGiovanna J, Nguyen TA, Micera S, Stokroos R, Kingma H, Guyot JP, Perez Fornos A. Vestibular implants: Hope for improving the quality of life of patients with bilateral vestibular loss. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:7192-5. doi: 10.1109/EMBC.2015.7320051. PMID 26737951
- [Background] Nguyen TA, DiGiovanna J, Cavuscens S, Ranieri M, Guinand N, van de Berg R, Carpaneto J, Kingma H, Guyot JP, Micera S, Fornos AP. Characterization of pulse amplitude and pulse rate modulation for a human vestibular implant during acute electrical stimulation. J Neural Eng. 2016 Aug;13(4):046023. doi: 10.1088/1741-2560/13/4/046023. Epub 2016 Jul 11. PMID 27396631
- [Background] DiGiovanna J, Nguyen TA, Guinand N, Perez-Fornos A, Micera S. Neural Network Model of Vestibular Nuclei Reaction to Onset of Vestibular Prosthetic Stimulation. Front Bioeng Biotechnol. 2016 Apr 20;4:34. doi: 10.3389/fbioe.2016.00034. eCollection 2016. PMID 27148528
- [Background] Guyot JP, Perez Fornos A, Guinand N, van de Berg R, Stokroos R, Kingma H. Vestibular assistance systems: promises and challenges. J Neurol. 2016 Apr;263 Suppl 1:S30-5. doi: 10.1007/s00415-015-7922-1. Epub 2016 Apr 15. PMID 27083882
- [Background] Guinand N, Van de Berg R, Cavuscens S, Stokroos R, Ranieri M, Pelizzone M, Kingma H, Guyot JP, Perez Fornos A. Restoring Visual Acuity in Dynamic Conditions with a Vestibular Implant. Front Neurosci. 2016 Dec 22;10:577. doi: 10.3389/fnins.2016.00577. eCollection 2016. PMID 28066163
- [Background] Nguyen TAK, Cavuscens S, Ranieri M, Schwarz K, Guinand N, van de Berg R, van den Boogert T, Lucieer F, van Hoof M, Guyot JP, Kingma H, Micera S, Perez Fornos A. Characterization of Cochlear, Vestibular and Cochlear-Vestibular Electrically Evoked Compound Action Potentials in Patients with a Vestibulo-Cochlear Implant. Front Neurosci. 2017 Nov 21;11:645. doi: 10.3389/fnins.2017.00645. eCollection 2017. PMID 29209162
- [Background] Guinand N, Van de Berg R, Cavuscens S, Ranieri M, Schneider E, Lucieer F, Kingma H, Guyot JP, Perez Fornos A. The Video Head Impulse Test to Assess the Efficacy of Vestibular Implants in Humans. Front Neurol. 2017 Nov 14;8:600. doi: 10.3389/fneur.2017.00600. eCollection 2017. PMID 29184530
- [Background] van de Berg R, Guinand N, Ranieri M, Cavuscens S, Khoa Nguyen TA, Guyot JP, Lucieer F, Starkov D, Kingma H, van Hoof M, Perez-Fornos A. The Vestibular Implant Input Interacts with Residual Natural Function. Front Neurol. 2017 Dec 14;8:644. doi: 10.3389/fneur.2017.00644. eCollection 2017. PMID 29312107
- [Background] Perez Fornos A, Cavuscens S, Ranieri M, van de Berg R, Stokroos R, Kingma H, Guyot JP, Guinand N. The vestibular implant: A probe in orbit around the human balance system. J Vestib Res. 2017;27(1):51-61. doi: 10.3233/VES-170604. PMID 28387690
- [Background] van de Berg R, Lucieer F, Guinand N, van Tongeren J, George E, Guyot JP, Kingma H, van Hoof M, Temel Y, van Overbeeke J, Perez-Fornos A, Stokroos R. The Vestibular Implant: Hearing Preservation during Intralabyrinthine Electrode Insertion-A Case Report. Front Neurol. 2017 Apr 10;8:137. doi: 10.3389/fneur.2017.00137. eCollection 2017. PMID 28443060
- [Background] Fornos AP, van de Berg R, Armand S, Cavuscens S, Ranieri M, Cretallaz C, Kingma H, Guyot JP, Guinand N. Cervical myogenic potentials and controlled postural responses elicited by a prototype vestibular implant. J Neurol. 2019 Sep;266(Suppl 1):33-41. doi: 10.1007/s00415-019-09491-x. Epub 2019 Aug 8. PMID 31396689
- [Background] Guyot JP, Perez Fornos A. Milestones in the development of a vestibular implant. Curr Opin Neurol. 2019 Feb;32(1):145-153. doi: 10.1097/WCO.0000000000000639. PMID 30566413
- [Background] Starkov D, Guinand N, Lucieer F, Ranieri M, Cavuscens S, Pleshkov M, Guyot JP, Kingma H, Ramat S, Perez-Fornos A, van de Berg R. Restoring the High-Frequency Dynamic Visual Acuity with a Vestibular Implant Prototype in Humans. Audiol Neurootol. 2020;25(1-2):91-95. doi: 10.1159/000503677. Epub 2019 Oct 29. PMID 31661687
- [Background] Seppen BF, van Hoof M, Stultiens JJA, van den Boogert T, Guinand N, Guyot JP, Kingma H, Fornos AP, Handschuh S, Glueckert R, Jacobi L, Schrott-Fischer A, Johnson Chacko L, van de Berg R. Drafting a Surgical Procedure Using a Computational Anatomy Driven Approach for Precise, Robust, and Safe Vestibular Neuroprosthesis Placement-When One Size Does Not Fit All. Otol Neurotol. 2019 Jun;40(5S Suppl 1):S51-S58. doi: 10.1097/MAO.0000000000002211. PMID 31225823
- [Background] Stultiens JJA, Postma AA, Guinand N, Perez Fornos A, Kingma H, van de Berg R. Vestibular Implantation and the Feasibility of Fluoroscopy-Guided Electrode Insertion. Otolaryngol Clin North Am. 2020 Feb;53(1):115-126. doi: 10.1016/j.otc.2019.09.006. Epub 2019 Oct 31. PMID 31677739
- [Background] Cretallaz C, Boutabla A, Cavuscens S, Ranieri M, Nguyen TAK, Kingma H, Van De Berg R, Guinand N, Perez Fornos A. Influence of systematic variations of the stimulation profile on responses evoked with a vestibular implant prototype in humans. J Neural Eng. 2020 Jun 12;17(3):036027. doi: 10.1088/1741-2552/ab8342. PMID 32213673
- [Background] van de Berg R, Ramos A, van Rompaey V, Bisdorff A, Perez-Fornos A, Rubinstein JT, Phillips JO, Strupp M, Della Santina CC, Guinand N. The vestibular implant: Opinion statement on implantation criteria for research. J Vestib Res. 2020;30(3):213-223. doi: 10.3233/VES-200701. PMID 32651339
- [Derived] van Boxel SCJ, Vermorken BL, Volpe B, Guinand N, Perez-Fornos A, Devocht EMJ, van de Berg R. Vestibular implant stimulation: pulse amplitude modulation versus combined pulse rate and amplitude modulation. J Neural Eng. 2025 Mar 28;22(2). doi: 10.1088/1741-2552/adc33a. PMID 40112351
- [Derived] Vermorken BL, van Boxel SCJ, Volpe B, Guinand N, Perez Fornos A, Devocht EMJ, van de Berg R. Rapid acclimatization to baseline stimulation with a multi-canal vestibulocochlear implant. Eur Arch Otorhinolaryngol. 2025 Jun;282(6):2991-3003. doi: 10.1007/s00405-024-09184-w. Epub 2025 Jan 30. PMID 39885011
- [Derived] Vermorken BL, Volpe B, van Boxel SCJ, Stultiens JJA, van Hoof M, Marcellis R, Loos E, van Soest A, McCrum C, Meijer K, Guinand N, Perez Fornos A, van Rompaey V, Devocht E, van de Berg R. The VertiGO! Trial protocol: A prospective, single-center, patient-blinded study to evaluate efficacy and safety of prolonged daily stimulation with a multichannel vestibulocochlear implant prototype in bilateral vestibulopathy patients. PLoS One. 2024 Mar 28;19(3):e0301032. doi: 10.1371/journal.pone.0301032. eCollection 2024. PMID 38547135
- See also: Related Info — http://www.vestibularimplant.com